CLINICAL TRIAL: NCT03333096
Title: Assessing Neurovisual Function in Patients With Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Ocuspecto Oy (Industry); European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: T212/2017
Record Dates: First submitted 2017-08-15; First posted 2017-11-06 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Glaucoma; Mild Cognitive Impairment; Glaucoma and Mild Cognitive Impairment; Healthy
Keywords: Glaucoma; Mild Cognitive Impairment; Ocusweep; Reaction Time; Neuropsychology; Dementia; Alzheimer's Disease; Brain Diseases
MeSH Terms: conditions — Glaucoma; Cognitive Dysfunction; Dementia; Alzheimer Disease; Brain Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glaucoma and mild cognitive impairment (Other): Device: Ocusweep test battery Neuropsychological test battery
  Ocusweep system compared to neuropsychological testing
  Interventions: Device: Ocusweep test battery; Diagnostic Test: Neuropsychological test battery

INTERVENTIONS:
Device: Ocusweep test battery — Ocusweep test battery to measure vision, visual system and cognitive performance including attention
  (Comparison of Ocusweep system to conventional neuropsychological test methods)
  (With the help of Ocusweep tests, information is obtained about the functioning of the whole visual system - from the ability of the eye to see to the efficiency of the brain to process visual information and the accuracy of eye movements)
Diagnostic Test: Neuropsychological test battery — Conventional neuropsychological test battery to measure executive functioning, attention, visuoconstructive abilities and processing speed

SUMMARY:
The aim of this study is to measure fitness to drive in patients with a visual and a cognitive impairment. To do so, Ocusweep is used in patients with glaucoma and Mild Cognitive Impairment. The participants will be divided over four groups; patients with glaucoma, patients with cognitive impairment, patients with both and a healthy control group. Differences in performance on Ocusweep in the four different groups of participants are expected. These effects may be related to fitness to drive, which is why those results will be compared to traditional neuropsychological measures of fitness to drive. the hypothesis of the current study is that the Ocusweep performance is related to performance on other measures of fitness to drive.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 65 years old
* Fit into one of the four groups of participants
* No other eye diseases than glaucoma
* Still be able to and allowed to drive a car
* Be able to visit the Turku Driver's Clinic for testing

Exclusion Criteria:

* A history of neurological disorders, depression or anxiety
* Motor problems
* Visual acuity less than 0.5
* Score over 6 in Geriatric Depression Scale questionnaire (GDS 15)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Perception speed | 2 years
  Measured by Ocusweep RTP-test
Evidence of cognitive impairment measured by MoCA-test | 2 years
  Measured with Montreal Cognitive Assessment. Outcome measure is a score between 0 and 30.
Evidence of impaired attentional ability - Cognitive profile | 2 years
  Measured by performing mazes. Unit of measure is seconds it takes to perform and number of errors.
Evidence of impaired Executive Functioning - Cognitive profile 1/2 | 2 years
  Measured by the Trail Making Test. Unit of measure is seconds to perform the test, which will be converted in a percentile score.
Evidence of impaired Executive Functioning - Cognitive profile 2/2 | 2 years
  Measured by the Trail Making Test. Unit of measure is errors made during the test.
Evidence of impaired Visuoconstructive abilities - Cognitive profile | 2 years
  Measured by the Benton Visual Retention Test. Unit of measure is number of correctly drawn designs (0-10)
Evidence of slow reaction time - Cognitive profile | 2 years
  Measured with Vienna Test System. Unit of measure is reaction time in ms. Results will be converted into percentile scores.
Evidence of impaired visual attention measured by UFOV-test - Cognitive Profile | 2 years
  Vision and visual attention measured with Useful Field of View. Unit of measure is milliseconds which is converted in group scores provided by UFOV.
Evidence of glaucomatous visual field defects 1/2 | 2 years
  Narrowing of the visual field measured with Standard Automated Perimetry (SAP).
Evidence of glaucomatous visual field defects 2/2 | 2 years
  Visual field defects measured by Ocusweep test called Reaction Time Perimetry. Outcome measure is reaction time on multiple locations on the visual field. From this data, unseen locations are calculated.
Contrast Sensitivity - Ocusweep | 2 years
  Evidence that Ocusweep finds patients not meeting health criteria for driving, measured by contrast sensitivity score.
Visual Acuity- Ocusweep | 2 years
  Evidence that Ocusweep finds patients not meeting health criteria for driving, measured by visual acuity score.
Visual Search - Ocusweep Neural | 2 years
  Measured in reaction time
Memory guided saccades - Ocusweep Neural | 2 years
  Measured in reaction time
Anti-saccades - Ocusweep Neural | 2 years
  Measured in reaction time
Prosaccade - Ocusweep Neural | 2 years
  Measured in reaction time

CONTACTS AND LOCATIONS:
Overall Officials: Eija Vesti, Dr, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland